CLINICAL TRIAL: NCT07132112
Title: A Single-arm, Open-label Clinical Study of GT719 Injection for Moderate to Severe Refractory Autoimmune Disease
Brief Title: GT719 Injection for Moderate to Severe Refractory Autoimmune Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-003-058
Record Dates: First submitted 2025-08-14; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Auto Immune Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: GT719 Injection

INTERVENTIONS:
Biological: GT719 Injection — GT719 Injection

SUMMARY:
This study is a prospective single-arm open-label clinical trial, including dose escalation and expansion phase, aims to evaluate the safety, efficacy, and cellular pharmacokinetics of GT719 Injection in patients with moderate to severe refractory autoimmune disease. A total of 30 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily enrolled in the study, signed an informed consent form, willing and able to comply with the study protocol.
* 2. Aged 18 to 65 years (inclusive), regardless of gender.

Specific inclusion criteria:

* 3. Participants with systemic lupus erythematosus (SLE)

  1. Meets the classification criteria for SLE in the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR);
  2. Disease activity score SLEDAI-2000 ≥ 6, with at least one British Islet Lupus Assessment Group Index (BILAG-2004) Grade A (severe manifestations) or two Grade B (moderate manifestations) organ scores, or both; Or the disease activity score SLEDAI-2000 ≥ 8;
* 4. Participants with idiopathic inflammatory myopathy （IIM）

  1. Complies with the 2017 EULAR/ACR classification criteria for inflammatory myopathy (including DM, PM, ASS, and NM)
  2. Myositis antibody positive;
  3. . Meets the definition of recurrence, refractory or progressive;
* 5. Participants with systemic sclerosis

  1. . Meet the 2013 American College of Rheumatology (ACR) SSc criteria;
  2. . SSc related antibodies are positive;
  3. . Meets the definition of refractory or progressive recurrence

Exclusion Criteria:

* 1. Within 3 weeks prior to lymphodepleting chemotherapy, complement inhibition therapy (such as Ecuzumab) has been used;
* 2. Received attenuated live vaccine within 4 weeks before lymphodepleting chemotherapy;
* 3. Having undergone major surgery within the 8 weeks prior to screening, or planning to undergo surgery during the study period;
* 4. Medical history of organ transplantation;
* 5. Previously received CAR-T product therapy targeting any target (excluding GT719 therapy);
* 6. According to the investigator's judgment, the situations that hinder participants from participating in the entire trial, confound the trial results, or participate in the trial that are not in the best interests of the participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing dose limiting toxicity | 28 days
  Proportion of participants experiencing dose limiting toxicity (DLT) within 28 days after cell infusion
Incidence of treatment-emergent adverse events | 2 years
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards

SECONDARY OUTCOMES:
Efficacy outcomes for SLE | 14 days; 1, 2, 3 and 6 Months post GT719 infusion
  SLE response index 4 (SR-4) response
Efficacy outcomes for Systemic Sclerosis | 14 days; 1, 2, 3, and 6 months post GT719 infusion
  ACR-CRISS score (CRISS score≥0.6 improvment, <0.6 no improvment)
Efficacy outcomes for Inflammatory Myopathy | 14 days; 1, 2, 3, and 6 months post GT719 infusion
  Total Improvement Score (TIS)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No